CLINICAL TRIAL: NCT01501747
Title: The Placebo Effect May Involve Modulating Drug Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: RAC2101105
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Placebo Effect; Drug Half Life; Pharmacokinetics
Keywords: Placebo effect; drug half life; pharmacokinetics
MeSH Terms: interventions — Caffeine; Acetaminophen; Cephalexin; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- overt drug (Active Comparator): The study has 4 sub-parts (one for each of 4 drugs), each sub-part has a crossover design. In this arm, the volunteer will be given one oral dose of 300 mg caffeine, 500 mg paracetamol, 500 mg cephalexin, or 400 mg ibuprofen and will be told that they are receiving such medication.
  Interventions: Drug: Caffeine, paracetamol, cephalexin, or ibuprofen
- Placebo (Covert drug) (Placebo Comparator): The study has 4 sub-parts (one for each of 4 drugs), each sub-part has a crossover design. In this arm, the volunteer will be given one oral dose of 300 mg caffeine, 500 mg paracetamol, 500 mg cephalexin, or 400 mg ibuprofen and will be told that they are receiving a placebo.
  Interventions: Drug: Placebo (caffeine, paracetamol, cephalexin, or ibuprofen)

INTERVENTIONS:
Drug: Caffeine, paracetamol, cephalexin, or ibuprofen — The study has 4 sub-parts (one for each of 4 drugs), each sub-part has a crossover design. In this arm, the volunteer will be given one oral dose of 300 mg caffeine, 500 mg paracetamol, 500 mg cephalexin, or 400 mg ibuprofen and will be told that they are receiving the active drug.
  Arms: overt drug
Drug: Placebo (caffeine, paracetamol, cephalexin, or ibuprofen) — The study has 4 sub-parts (one for each of 4 drugs), each sub-part has a crossover design. In this arm, the volunteer will be given one oral dose of 300 mg caffeine, 500 mg paracetamol, 500 mg cephalexin, or 400 mg ibuprofen and will be told that they are receiving a placebo.
  Arms: Placebo (Covert drug)

SUMMARY:
The total effect of a medication is the sum of its drug effect, placebo effect (meaning response of placebo), and their interaction. Current interpretation of clinical trials (the gold standard of evidence-based-medicine) assumes no interaction, and the mechanism(s) underlying such interaction have not been fully explored. One possibility is that the placebo effect may modulate drug bioavailability. Using caffeine as a model drug, we have recently shown that the placebo effect of caffeine ingestion prolongs caffeine half life. Due to the novelty of this finding and its important clinical practice and clinical research implications, it needs to be confirmed in another set of subjects and extended to additional drugs.

The results of the study are expected to further our understanding of the mechanism of action of a widely used medical intervention, i.e., placebo. The results will be important for both clinical practice and clinical research.

DETAILED DESCRIPTION:
The total effect of a medication is the sum of its drug effect, placebo effect (meaning response of placebo), and their interaction. Current interpretation of clinical trials (the gold standard of evidence-based-medicine) assumes no interaction, and the mechanism(s) underlying such interaction have not been fully explored. One possibility is that the placebo effect may modulate drug bioavailability. Using caffeine as a model drug, we have recently shown that the placebo effect of caffeine ingestion prolongs caffeine half life. Due to the novelty of this finding and its important clinical practice and clinical research implications, it needs to be confirmed in another set of subjects and extended to additional drugs.

DESIGN: Balanced cross-over, single-dose, two-period, two-group deign comparing caffeine, paracetamol, cephalexin, and ibuprofen described as such (overt) to the same medication described as placebo (covert).

METHODS: 32, 50, 50, and 30 healthy adult volunteers will be enrolled in the caffeine (300 mg), paracetamol (500 mg), cephalexin (500 mg), and ibuprofen (400 mg) cross-over studies, respectively. Volunteers will be partially deceived to the intervention assignment (i.e., in the covert arm). Serum levels of each drug will be blindly determined by locally validated HPLC assays. Plasma half life (primary outcome) as well as Cmax, Tmax, and AUC (secondary outcomes) of each drug will be determined and analyzed by ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Having no evidence of clinically important deviation from normal health as indicated by medical history, vital signs, and clinical laboratory tests.
* Acceptance to abstain from taking any medication other than birth control pills (including over-the-counter drugs) for at least 1 week prior to, and during the study; and from smoking and taking alcohol or caffeine or related xanthenes-containing beverages or food for 48 hours before and throughout each study period.
* Having good peripheral venous access.
* For the caffeine study, habitual daily caffeine intake should be 100-300 mg.

Exclusion Criteria:

* Women should be non-pregnant and non-lactating. For menstruating women, the study will be conducted 5 to 19 days after the last menstrual period and a urine pregnancy test will be performed.
* Should not have history of hypersensitivity to the drug to be tested or to its related compounds.
* Body Mass Index (BMI) should be less than 35 kg/m2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Plasma half life | 24 hours
  The study has 4 sub-parts (one for eah of 4 drugs), each sub-part has a crossover design. The time frame to measure the outcome depends on the drug studied. For caffeine it is 24 hours, for paracetamol, it is 14 hours, for cephalexin, it is 6 hours, and for ibuprofen, it is 10 hours.

SECONDARY OUTCOMES:
Area under the curve | 24 hours
  The study has 4 sub-parts (one for eah of 4 drugs), each sub-part has a crossover design. The time frame to measure the outcome depends on the drug studied. For caffeine it is 24 hours, for paracetamol, it is 14 hours, for cephalexin, it is 6 hours, and for ibuprofen, it is 10 hours.
Tmax | 24 hours
  The study has 4 sub-parts (one for eah of 4 drugs), each sub-part has a crossover design. The time frame to measure the outcome depends on the drug studied. For caffeine it is 24 hours, for paracetamol, it is 14 hours, for cephalexin, it is 6 hours, and for ibuprofen, it is 10 hours.
Cmax | 24 hours
  The study has 4 sub-parts (one for eah of 4 drugs), each sub-part has a crossover design. The time frame to measure the outcome depends on the drug studied. For caffeine it is 24 hours, for paracetamol, it is 14 hours, for cephalexin, it is 6 hours, and for ibuprofen, it is 10 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Hammami MM, Yusuf A, Shire FS, Hussein R, Al-Swayeh R. Does the placebo effect modulate drug bioavailability? Randomized cross-over studies of three drugs. J Negat Results Biomed. 2017 May 23;16(1):10. doi: 10.1186/s12952-017-0075-2. PMID 28535819